CLINICAL TRIAL: NCT04855968
Title: The Effect of Mindfulness/Meditation on Post-operative Pain and Opioid Consumption
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient compliance
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, MD, Principal investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000950
Record Dates: First submitted 2021-02-02; First posted 2021-04-22 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Tears
Keywords: Shoulder Arthroscopy; head space; mindfulness; Subacromial bursitis; biceps tenodesis
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (CON) (Active Comparator): will receive the usual standard of care post-operative pain pills for the involved shoulder (Control Group)
  Interventions: Other: Patients will take standard post-op pain medication
- Mindfulness/Meditation (MM) (Experimental): will receive the usual standard of care post-operative pain pills for the involved shoulder with the addition of access to the Headspace application for mindfulness/meditation (Mindfulness/Meditation Group)
  Interventions: Other: In addition to standard post-op medication patient will have access to the head space meditation application.

INTERVENTIONS:
Other: In addition to standard post-op medication patient will have access to the head space meditation application. — Patients will receive access to head space meditation application in addition to standard pain medication post surgery.
  Arms: Mindfulness/Meditation (MM)
Other: Patients will take standard post-op pain medication — Standard post-op pain medication
  Arms: control (CON)

SUMMARY:
The objective of this study is to examine the effectiveness of mindfulness/meditation using the Headspace App on post-operative pain and opioid consumption in patients after arthroscopic rotator cuff repairs, biceps tenodesis, and Mumford procedures.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of mindfulness/meditation on post-operative pain and opioid consumption. Patients will be randomized into one of two standardized groups after shoulder arthroscopy: Control group (CON) and mindfulness/meditation group (MM). All participants will be consented and enrolled into the study before surgery. Both groups will receive the same standardized method of post-operative pain medication for post-operative pain relief. Participants in the MM group will utilize a Headspace application on their smart phone meditate twice a day while the control group will not perform any meditation or mindfulness. Patient reported outcomes will be collected at regular intervals. Patients age 18 and older undergoing shoulder arthroscopy for rotator cuff repair and/or biceps tenodesis and/or Mumford procedure. The study includes 3 visits which are standard of care pre-operative and post-operative visits. The duration of the study will be 6 months which will include 3 standard of care post-operative visits and electronic surveys to track patient reported outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Status post shoulder arthroscopy for rotator cuff repair, biceps tendinopathy, and/or Mumford Procedure

Exclusion Criteria:

* Less than 18 years old
* Patients undergoing a simultaneous arthroscopic procedure that is not in the inclusion criteria.
* History of shoulder osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 2 weeks post-op
  single-item measure of pain and consists of a 100 millimeter (mm) horizontal line with the labels "No Pain" at the leftmost portion and "Worst Pain" at the rightmost portion of the line
visual analog scale | 6 weeks post-op, 3months post-op and 6 months post-op
  single-item measure of pain and consists of a 100 millimeter (mm) horizontal line with the labels "No Pain" at the leftmost portion and "Worst Pain" at the rightmost portion of the line
visual analog scale | 3months post-op
  single-item measure of pain and consists of a 100 millimeter (mm) horizontal line with the labels "No Pain" at the leftmost portion and "Worst Pain" at the rightmost portion of the line
visual analog scale | 6 months post-op
  single-item measure of pain and consists of a 100 millimeter (mm) horizontal line with the labels "No Pain" at the leftmost portion and "Worst Pain" at the rightmost portion of the line
number of opioid pills | 2 weeks post-op
  number of pills taken at each time point
number of opioid pills | 6 weeks post-op
  number of pills taken at each time point
number of opioid pills | 3 months post-op
  number of pills taken at each time point
number of opioid pills | 6months post-op
  number of pills taken at each time point

SECONDARY OUTCOMES:
compliance of the intervention in the MM groups which will be tracked via the Headspace application. | 2 weeks post-op
  used to detect the association between using the Headspace application and the amount of post-operative pain
compliance of the intervention in the MM groups which will be tracked via the Headspace application. | 6 weeks post-op
  used to detect the association between using the Headspace application and the amount of post-operative pain
compliance of the intervention in the MM groups which will be tracked via the Headspace application. | 3 months post-op
  used to detect the association between using the Headspace application and the amount of post-operative pain
compliance of the intervention in the MM groups which will be tracked via the Headspace application. | 6 months post-op
  used to detect the association between using the Headspace application and the amount of post-operative pain
Patient reported out comes :Single Assessment Numeric Evaluation (SANE) | 2 weeks post-op
  composed of a single question, would be a valid and responsive instrument to provide a global assessment of patients shoulder function on a scale of 1-100
Patient reported out comes :Single Assessment Numeric Evaluation (SANE) | 6 weeks post-op
  composed of a single question, would be a valid and responsive instrument to provide a global assessment of patients shoulder function on a scale of 1-100
Patient reported out comes :Single Assessment Numeric Evaluation (SANE) | 3 months post-op
  composed of a single question, would be a valid and responsive instrument to provide a global assessment of patients shoulder function on a scale of 1-100
Patient reported out comes :Single Assessment Numeric Evaluation (SANE) | 6 moths post-op.
  composed of a single question, would be a valid and responsive instrument to provide a global assessment of patients shoulder function on a scale of 1-100
Patient reported out comes: The Veterans RAND 12 Item Health Survey (VR-12) | 2 weeks post-op.
  12 question ,patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Patient reported out comes: The Veterans RAND 12 Item Health Survey (VR-12) | 6 weeks post-op.
  12 question ,patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Patient reported out comes: The Veterans RAND 12 Item Health Survey (VR-12) | 3 months post-op.
  12 question ,patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Patient reported out comes: The Veterans RAND 12 Item Health Survey (VR-12) | 6 months post-op.
  12 question ,patient-reported global health measure that is used to assess a patient's overall perspective of their health.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Banffy, MD, Principal Investigator — Cedar Sinai -Kerlan Jobe
Locations (1):
- Kerlan Jobe, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No